CLINICAL TRIAL: NCT02213029
Title: Study IVF116828:A Multi-Cohort Phase I Study to Investigate the Pharmacokinetics, Pharmacodynamics and Tissue Concentrations of Epelsiban (GSK557296) in Healthy Female Volunteers During Control and Challenge States With and Without Oxytocin
Brief Title: A Study to Evaluate Pharmacokinetics, Pharmacodynamics and Tissue Concentrations of Epelsiban
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 116828
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Embryo Transfer
Keywords: epelsiban; pharmacokinetics; patient reported pain / discomfort; pharmacodynamics; oxytocin infusions; Uterine contractions
MeSH Terms: interventions — epelsiban; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oxytocin or Placebo challenge (Cohort 1) (Experimental): Subjects will receive oxytocin and or placebo challenges as escalating intravenous (IV) infusions administered on the day of ovulation, followed by an IV bolus day 1 post ovulation, and an intramuscular (IM) injection day 2 post ovulation. The planed doses and routes of administration of oxytocin are as follows: IV infusion will be initiated at 5 milliunit/minute (mU/min) and maintained for 60 min, then the rate will be increased to 10 mU/min and maintained for 60 minutes, a final escalation to 20mU/min will be maintained for 60 minutes, after which the infusion will be stopped. For the IV bolus, a single 5 International unit (IU) IV bolus will be administered. For the IM dosing, a single 10 IU IM injection will be administered.
  Interventions: Drug: Placebo; Drug: Oxytocin; Drug: Ortho-Cylcen (21)® tablet
- Epelsiban or Placebo (Cohort 2) (Experimental): Subjects in Cohort 2A will receive first dose of epelsiban (25mg) or placebo after receiving initial oxytocin challenge with dose selected in Cohort 1 followed by 30 minutes washout period. Subjects will receive second dose of epelsiban (150mg) or placebo 12 hours after first dose. Based on the results of Cohort 2A, additional doses may be investigated with a new Cohort 2B (<150mg) and Cohort 2C (>200mg) with repeated oxytocin challenges.
  Interventions: Drug: Epelsiban; Drug: Placebo; Drug: Oxytocin; Drug: Ortho-Cylcen (21)® tablet
- Biopsy cohort (Cohort 3) (Experimental): Subjects will receive first dose of epelsiban 150mg without oxytocin challenge followed by second dose of epelsiban 150mg 24 hours after the first dose. Subsequently one hour after the second dose, subjects will undergo endometrial biopsies.
  Interventions: Drug: Epelsiban; Drug: Ortho-Cylcen (21)® tablet

INTERVENTIONS:
Drug: Epelsiban — White to off white Oral tablets with unit dose strength of 5 mg or 25 mg for dose level of 25 mg, 150mg or >150mg
  Arms: Biopsy cohort (Cohort 3); Epelsiban or Placebo (Cohort 2)
Drug: Placebo — White to off white oral placebo tablets to match 5mg epelsiban
  Arms: Epelsiban or Placebo (Cohort 2); Oxytocin or Placebo challenge (Cohort 1)
Drug: Oxytocin — Oxytocin for IV infusion (at doses of 5, 10, and 20 milliunits), IV bolus (5 IU administered IV as a bolus over 15 seconds) and IM (5 IU administered IM).
  Arms: Epelsiban or Placebo (Cohort 2); Oxytocin or Placebo challenge (Cohort 1)
Drug: Ortho-Cylcen (21)® tablet — White, blue or green tablets for oral administration per product insert to synchronize the menstrual cycles with ovulation. Ortho Cyclen (21) ® is a registered trademark of Johnson & Johnson

SUMMARY:
This multi-cohort phase I study is designed to assess the pharmacokinetics (PK) and pharmacodynamics (PD) of oxytocin and to evaluate epelsiban (GSK557296) potential to reduce subendometrial contractractility induced by oxytocin in healthy female subjects. Additionally tissues concentrations of epelsiban will be determined from endometrial tissue biopsies. Data from this study will inform the identification of the doses of epelsiban to be used in future in-vitro fertilization (IVF) clinical studies. Expected number of subjects to be randomized are: Cohort 1- 10 subjects, Cohort 2a- 10 subjects for each epelsiban arm 25 milligrams (mg), 200mg, 5 for placebo, Cohort 2b- 10 subjects per arm with dose to be determined, cohort 3- 6 subjects. Cohorts 1 and 2 will be double blind (sponsor unblinded) placebo controlled cohorts. Cohort 3 will be an open label cohort, cohort 4 will be a double blind (sponsor unblinded) placebo controlled cohort.

ELIGIBILITY:
Inclusion Criteria:

For ultrasound training cohort

* Female volunteers of childbearing potential; with a negative pregnancy test as determined by human chorionic gonadotropin (hCG) testing at screening and prior to study initiation.
* Age between 18 and 35 years old (inclusive).
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 18-30 kg/meter (m)^2 (inclusive).
* Normal ovarian and uterine anatomy as assessed by transvaginal ultrasonography.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Is in good physical and mental health as determined by a responsible and experienced physician, based on a medical evaluation including medical history, and physical examination.

For Cohorts 1, 2A, 2B, 2C, 3

* Female volunteers of childbearing potential; with a negative pregnancy test as determined by hCG testing at screening and prior to study initiation.
* Agrees to use one of the contraception methods for 2 weeks prior to the start of study to minimize the risk of pregnancy. Female subjects must agree to use contraception until at least 48 hours have passed after the last dose of study drug. OR has only same-sex partners, when this is her preferred and usual lifestyle. Oral contraceptive (OC) pill naive or have discontinued OC at least 2 months prior to study entry.
* Age between 18 and 35 years old.
* Body weight >=50 kg and BMI within the range 18-30 kg/m^2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form as signed consent form; and is in good physical and mental health as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GlaxoSmithKline (GSK) Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Subjects with a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli international unit (MI)U/milliliter (mL) and estradiol <40 picogram/mL (<147 picomoles/Liter) should always be excluded from enrolment.
* based on single or averaged corrected QTc values of triplicate ECGs obtained over a brief recording period: QTc <450 milliseconds (msec); or QTc <480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

For Training Cohort

* Ultrasonographic evidence of uterine anomalies, including but not limited to intramural or submucosal leiomyomas (fibroids) cysts, endometrial polyps, American Society for Reproductive Medicine (ASRM) Class I-VI uterine malformations or intrauterine fluid collections.
* Pregnancy (suspected or diagnosed) or lactation.
* Has had a prior partial or total hysterectomy or tubal ligation.
* Currently using and intrauterine device (IUD) for any reason.
* History or suspicion of drug or alcohol abuse. Criteria Based Upon Medical Histories For Training Cohort
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >7 drinks. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.

Criteria Based Upon Diagnostic Assessments For Training Cohort

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive pre-study drug/alcohol/; and.
* A positive test for human immune virus (HIV) antibody. For Cohorts 1, 2A, 2B, 2C, 3
* Female with an abnormal obstetric profile (average durations <27 days or > 31 days;Any contraindication for oral contraception use; Is using hormone replacement therapy (HRT); Ultrasonographic evidence of ovarian dysfunction, such as Polycystic Ovary Syndrome (PCOS) or ovarian anomalies such as dermoid or hemorrhagic cysts; Ultrasonographic evidence of uterine anomalies, including but not limited to intramural or submucosal leiomyomas (fibroids) cysts, endometrial polyps, ASRM Class I-VI uterine malformations or intrauterine fluid collections.
* Pregnancy (suspected or diagnosed) or lactation.
* Has had a prior partial or total hysterectomy or tubal ligation.
* Has had prior surgical procedures to the cervix (cryoablation, loop electrical excision procedure [LEEP] or other similar procedures).
* Currently using an IUD for any reason.
* Potential volunteers who are at high risk of developing complications while taking oral contraceptives will not be entered into the study in accordance with normal standards of good clinical practice.
* History or suspicion of drug or alcohol abuse. Criteria Based Upon Medical Histories For Cohorts 1, 2, 3
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >7 drinks. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of hypertension, use of an anti-hypertensive, or any systolic blood pressure >=140 millimeter of mercury (mmHg) or diastolic blood pressure >=90 mmHg.

Criteria Based Upon Diagnostic Assessments For Cohorts 1, 2, 3

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive pre-study drug/alcohol/cotinine screen.
* A positive test for HIV antibody. Other Criteria
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2016-02-07 (Actual); Study Completion 2016-02-07 (Actual)

PRIMARY OUTCOMES:
The effect of the infused oxytocin dose on the time course of the frequency of endometrial contractions in Cohort 1 during the periovulatory phase | Up to Day 3
  The relationship between the dose of the infused oxytocin and the time course of the frequency of endometrial contractions in Cohort 1 during the periovulatory phase (ovulation to 3-5 days post ovulation) will be assessed to establish the PD response from the oxytocin infusions and endometrial contraction rate which will provide the oxytocin infusion challenge dose to use in Cohort 2. If data permit, the effective dose 50 (ED50) of oxytocin will be also be determined. Uterine contraction rates, contractility measures, etc. will be measured by computer assisted ultrasound image analyses.
Frequency of endometrial contractions in Cohorts 2A, 2B and 2C during the periovulatory phase and 3-5 days post ovulation. | Up to Day 2
  Frequency of endometrial contractions will be assessed to evaluate the dose response relationship for epelsiban with respect to its ability to reduce endometrial contractions in the study population exposed to repeated oxytocin challenges. Uterine contraction rates, contractility measures, etc. will be measured by computer assisted ultrasound image analyses.
Reduction in the frequency of subendometrial contractions in Cohorts 2 A, B and C, all during the periovulatory phase. | Up to Day 2
  The reduction in the frequency of subendometrial contractions will be assessed during the periovulatory phase to investigate the PD response of epelsiban in the study population when exposed to repeated oxytocin challenges. If data permit, the infectious dose 50 (ID50) of epelsiban will also be determined. Uterine contraction rates, contractility measures, etc. will be measured by computer assisted ultrasound image analyses.
The duration of the reduction in subendometrial contractions in Cohorts 2 A, B and C, all during the periovulatory phase | Up to Day 2
  The duration of the reduction in subendometrial contractions will be assessed during the periovulatory phase to investigate the PD response of epelsiban in the study population when exposed to repeated oxytocin challenges. If data permit, the infectious dose 50 (ID50) of epelsiban will also be determined. Uterine contraction rates, contractility measures, etc. will be measured by computer assisted ultrasound image analyses.
Plasma concentrations of epelsiban or metabolite and the reduction of subendometrial contraction frequency in Cohorts 2 A, B and C, all during the periovulatory phase. | PK samples will be collected at 3, 3.25, 3.5, 4, 6.5, 11, 15, 27, 31 and 39 hours post dose in cohort 2.
  The relationship between the plasma concentrations and the reduction of subendometrial contraction frequency will be assessed during the periovulatory phase to establish the PK/PD relationship between epelsiban (and/or its metabolites) and endometrial contraction rate in the study population exposed to repeated oxytocin challenges. If data permit, the maximum inhibitory effect (Imax) and IC50 of epelsiban will also be determined. Uterine contraction rates, contractility measures, etc. will be measured by computer assisted ultrasound image analyses.

SECONDARY OUTCOMES:
Frequency of endometrial and subendometrial contractility in Cohort 2. | Up to Day 3
  Following parameters will be assessed: Wave period, external contractile measure, internal contractile measure and total contractile measure, wave directionality, wave amplitude and wave completeness.
Frequency of subendometrial contractility in Cohort 3 | Up to Day 2
  To evaluate the endometrial and subendometrial contractions following epelsiban dose in the absence of oxytocin challenges.
Number of subjects with adverse events in Cohort 1 | 18 days
  AEs will be collected from the start of Study Treatment and until the follow-up contact.
Number of subjects with adverse events (AEs) in Cohort 2 | 17 days
  AEs will be collected from the start of Study Treatment and until the follow-up contact.
Number of subjects with adverse events in Cohort 3 | 16 days
  AEs will be collected from the start of Study Treatment and until the follow-up contact.
Change from Baseline in laboratory parameters in Cohort 1 | Baseline (screening) and upto 21 days
  Laboratory parameters include: hematology, clinical chemistry, urinalysis
Change from Baseline in laboratory parameters in Cohort 2 | Baseline (screening) and upto 20 days
  Laboratory parameters include: hematology, clinical chemistry, urinalysis
Change from Baseline in laboratory parameters Cohort 3 | Baseline (screening) and upto 19 days
  Laboratory parameters include: hematology, clinical chemistry, urinalysis
Change from Baseline in vital signs in Cohort 1 | Baseline (screening) and upto 21 days
  Vital signs measurement include: blood pressure, pulse pressure, heart rate.
Change from Baseline in vital signs in Cohort 2 | Baseline (screening) and upto 20 days
  Vital signs measurement include: blood pressure, pulse pressure, heart rate.
Change from Baseline in vital signs in Cohort 3 | Baseline (screening) and upto 19 days
  Vital signs measurement include: blood pressure, pulse pressure, heart rate.
Change from Baseline in electrocardiogram (ECG) parameters in Cohort 1 | Baseline (screening) and upto 21 days
  ECG parameters include: PR, QRS, QT, and corrected QT (QTc) intervals.
Change from Baseline in ECG parameters in Cohort 2 | Baseline (screening) and upto 20 days
  ECG parameters include: PR, QRS, QT, and corrected QT (QTc) intervals.
Change from Baseline in ECG parameters in Cohort 3 | Baseline (screening) and upto 19 days
  ECG parameters include: PR, QRS, QT, and corrected QT (QTc) intervals.
Composite of PK parameters following epelsiban dosing | PK samples will be collected at 3, 3.25, 3.5, 4, 6.5, 11, 15, 27, 31 and 39 hours post dose in cohort 2.
  PK parameters will be assessed for epelsiban and its metabolite (GSK2395448). PK parameters include: maximum plasma concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve (AUC), apparent terminal phase half-life (t1/2), renal clearance (CL).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, Baltimore, Maryland

REFERENCES:
- See also: Results for study 116828 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116828?search=study&b'search_terms=116828'#rs